CLINICAL TRIAL: NCT00387322
Title: Phase I/II Study of Two Different Schedules of Pemetrexed (ALIMTA) and Erlotinib (TARCEVA) in Advanced Solid Tumors, With Emphasis on Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pemetrexed Disodium and Erlotinib in Treating Patients With Advanced Non-Small Cell Lung Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: David Gandara, MD, University of California Davis Cancer Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000505895; P30CA093373 (NIH); UCDCC-159 (Other: University of California, Davis - Cancer Center); 200412741 (Other: University of California, Davis - IRB)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients receive oral erlotinib hydrochloride once on days 2, 9, and 16 and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of unacceptable toxicity or disease progression
  Interventions: Drug: erlotinib hydrochloride; Drug: pemetrexed disodium
- Group 2 (Experimental): Patients receive oral erlotinib hydrochloride once daily on days 2-16 and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: erlotinib hydrochloride; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: Tarceva
Drug: pemetrexed disodium — Given IV
  Other Names: Alimta

SUMMARY:
RATIONALE: Pemetrexed disodium and erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pemetrexed disodium together with erlotinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of two different schedules of pemetrexed disodium and erlotinib and to see how well they work in treating patients with advanced non-small cell lung cancer or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of combining pemetrexed disodium with erlotinib hydrochloride in patients with advanced non-small lung cancer (NSCLC) or other solid tumors. (Phase I)
* Determine the response rate in patients with NSCLC treated with pemetrexed disodium in combination with erlotinib hydrochloride. (Phase II)

Secondary

* Compare toxicity differences between different schedules of pemetrexed disodium and erlotinib hydrochloride. (Phase I)
* Determine the maximum tolerated dose (MTD) of 2 different schedules of pemetrexed disodium and erlotinib hydrochloride. (Phase I)
* Determine, preliminarily, the efficacy of the combination of pemetrexed disodium and erlotinib hydrochloride in patients with advanced solid tumors. (Phase I)
* Assess the overall survival and progression-free survival. (Phase II)
* Determine the frequency and severity of toxicities associated with the administration of pemetrexed disodium and erlotinib hydrochloride. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study followed by a phase II open-label study.

* Phase I: Patients are assigned to 1 of 2 treatment groups in an alternating fashion. Once accrual to the first dose level in group 1 is complete, group 2 will open for accrual to its first dose level.

  * Group 1: Patients receive oral erlotinib hydrochloride once on days 2, 9, and 16 and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of unacceptable toxicity or disease progression.
  * Group 2: Patients receive oral erlotinib hydrochloride once daily on days 2-16 and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of unacceptable toxicity or disease progression.

In both groups, patients may continue to receive erlotinib hydrochloride alone after completion of 6 courses of erlotinib hydrochloride in combination with pemetrexed disodium.

In both groups, cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride and pemetrexed disodium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive pemetrexed disodium at the MTD and erlotinib hydrochloride at the MTD as in group 1 or 2 (whichever is more favorable).

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 92 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* For the phase I portion of the study patients must have cytologically or histologically proven advanced solid tumors for which there is no standard effective therapy available. For the phase II portion patients must have cytologically or histologically proven selected stage IIIB (pleural effusion) or IV NSCLC. Patients with NSCLC that have progressed or recurred after first-line therapy for stage IIIA or IIIB may also be considered.
* For the phase II portion patients must have disease that has progressed or recurred after treatment with platinum-based therapy.
* Any number of prior chemotherapy regimens are allowed for the phase I portion and no more than 1 previous treatment for advanced NSCLC is allowed for the phase II portion.
* Patients must have measurable disease by RECIST criteria. Disease in previously irradiated sites is considered measurable if there is clear disease progression following radiation therapy. Patients with evaluable disease (bone metastases, pleural fluid, ascites, etc.) may be included in the phase I portion of the trial.
* Patients must be 18 years of age or older.
* Patients must have a performance status of 0-2 for phase I portion of study and a performance status of 0 -1 for the phase II portion of the trial.
* Patients must have an estimated survival of at least 3 months.
* Any prior chemotherapy that patients have received has to have been completed at least 4 weeks prior to start of treatment. For prior mitomycin chemotherapy a 6-week interval is required. Prior radiation must have been completed at least 2 weeks prior to start of therapy. Patients must have recovered from acute reversible side effects of prior chemotherapy regimens or radiotherapy to NCI-CTC < grade 1 (excluding alopecia).
* Patients must have adequate renal function as documented by a serum creatinine < 1.5 mg/dl or a calculated creatinine clearance of > 45 ml/min (see appendix for formula for calculating creatinine clearance).
* Patients must have adequate liver function as documented by serum bilirubin < 1.5 x ULN. AST must be < 2.5 x institutional upper limit of normal.
* Patients must have a pretreatment granulocyte count of >1500/mm3 and platelet count of >100 000/mm3.
* Patients with asymptomatic treated brain metastasis (surgical resection or radiotherapy) may be included if they are neurologically stable and have been off steroids and anticonvulsants for at least 4 weeks. Because of the possibility of treatment related neurological toxicity it is difficult to evaluate for toxicity in the presence of symptomatic brain metastasis.
* All patients must give voluntary written informed consent.
* Patients must be able to take and retain oral medication.
* Patients of reproductive potential must agree to use effective contraceptive method while on treatment and for 3 months afterwards as the effects of these drugs on the unborn fetus are unknown.
* Patients on coumadin should have their INR monitored at least once per week or more frequently depending on the investigators judgement. There have been some case reports of increased INR when coumadin is co-administered with OSI-774/placebo.

Exclusion Criteria:

* Patients may not have previously received Pemetrexed or an EGFR-directed therapy.
* Females can not be pregnant or breastfeeding as the effects of these drugs on the unborn fetus are unknown. Documentation of a negative serum pregnancy test is required for all women of reproductive potential.
* Patients with symptomatic brain metastasis or still requiring steroids and anti-convulsants may not be included.
* No other prior malignancy is allowed for the phase II portion except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for over five years.
* Patients cannot take non-steroidal anti-inflammatory agents (NSAIDS) or salicylates 2 days prior and 2 days following (5 days pre and post for long-acting NSAIDS) administration of pemetrexed due to concerns of increased risk of renal toxicity.
* Patients with clinically significant ophthalmologic abnormalities will be excluded. This includes severe dry eye syndrome, keratoconjunctivitis sicca, Sjogren's syndrome, severe exposure keratopathy, or other disorders that might increase the risk of corneal epithelial injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-03; Primary Completion 2007-10 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility (Phase I) | October 2007
Response rate (Phase II) | Phase II not performed

SECONDARY OUTCOMES:
Toxicity (Phase I) | October 2007
Maximum tolerated dose (Phase I) | October 2007
Preliminary efficacy (Phase I) | October 2007
Overall survival (Phase II) | Phase II not performed
Progression-free survival (Phase II) | Phase II not performed
Frequency and severity of toxicity (Phase II) | Phase II not performed

CONTACTS AND LOCATIONS:
Overall Officials: David Gandara, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Result] Davies AM, Ho C, Beckett L, Lau D, Scudder SA, Lara PN, Perkins N, Gandara DR. Intermittent erlotinib in combination with pemetrexed: phase I schedules designed to achieve pharmacodynamic separation. J Thorac Oncol. 2009 Jul;4(7):862-8. doi: 10.1097/JTO.0b013e3181a94b08. PMID 19494788